CLINICAL TRIAL: NCT04501640
Title: A Phase 4 Open-label, Randomized, Single Oral Dose, Two-way Crossover Study to Investigate the Effect of Food on the Pharmacokinetics of Mirabegron in Healthy Chinese Subjects
Brief Title: A Study to Investigate the Effect of Food With Mirabegron in Healthy Chinese Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 178-MA-2294; CTR20201670 (Registry Identifier: ChinaDrugTrials.org.cn)
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Results first posted 2021-10-29 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Pharmacokinetics of Mirabegron; Food Effect; Healthy Chinese Subjects
Keywords: mirabegron; pharmacokinetics; two-way crossover
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: This was a two-way crossover design with 2 period and 2 dose groups. Participants were randomized to 1 of 4 sequences dependent on dose and period assigned.
Masking Description: This was an open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Mirabegron 25 mg fed/Mirabegron 25 mg fasted (Experimental): Participants received single dose of 25 mg mirabegron tablet under fed condition orally, on day 1 of period 1 followed by single dose of 25 milligram (mg) mirabegron tablet under fasted condition orally, on day 1 of period 2. A washout period of 10 days was maintained between the mirabegron administrations in each period.
  Interventions: Drug: mirabegron
- Mirabegron 25 mg fasted/Mirabegron 25 mg fed (Experimental): Participants received single dose of 25 mg mirabegron tablet under fasted condition orally, on day 1 of period 1 followed by single dose of 25 mg mirabegron tablet under fed condition orally, on day 1 of period 2. A washout period of 10 days was maintained between the mirabegron administrations in each period.
  Interventions: Drug: mirabegron
- Mirabegron 50 mg fed/Mirabegron 50 mg fasted (Experimental): Participants received single dose of 50 mg mirabegron tablet under fed condition orally, on day 1 of period 1 followed by single dose of 50 mg mirabegron tablet under fasted condition orally, on day 1 of period 2. A washout period of 10 days was maintained between the mirabegron administrations in each period.
  Interventions: Drug: mirabegron
- Mirabegron 50 mg fasted/Mirabegron 50 mg fed (Experimental): Participants received single dose of 50 mg mirabegron under fasted condition orally, on day 1 of period 1 followed by single dose of 50 mg mirabegron tablet under fed condition orally, on day 1 of period 2. A washout period of 10 days was maintained between the mirabegron administrations in each period.
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — Oral adminstration
  Other Names: Betmiga

SUMMARY:
This study determined the effect of food on the pharmacokinetics (PK) of single oral doses of mirabegron in healthy Chinese male and female participants.

This study also evaluated the safety and tolerability of single oral doses of mirabegron in healthy Chinese male and female participants.

DETAILED DESCRIPTION:
An open-label, randomized, 2-period, single oral dose crossover design at 2 dose levels in healthy Chinese male and female participants. Each participant took part in 2 periods separated by a washout of at least 10 days between investigational product (IP) administrations in each period.

Participants were screened for up to 21 days prior to IP administration on day 1 of period 1. Eligible participants were admitted to the clinical unit on day -1 of each period and were confined until the last pharmacokinetic sample had been drawn within each period. PK samples were collected predose on day 1 of each period and at multiple time points following each dose.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index range of 19.0 to 24.9 kg/m^2, inclusive and weighs at least 50 kg for male subjects and 45 kg for female subjects at screening.
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after final IP administration
* Female subject must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final IP administration.
* Female subject must not donate ova starting at first dose of IP and throughout the study period and for 30 days after final IP administration.
* Male subject with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the study period and for 30 days after final IP administration.
* Male subject must not donate sperm during the study period and for 30 days after final IP administration.
* Male subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after final IP administration.
* Subject agrees not to participate in another interventional study while participating in the present study, defined as 84 days prior screening until completion of the last study visit.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to mirabegron or any components of the formulation used.
* Subject has had previous exposure with mirabegron.
* Subject has any of the liver function tests (alkaline phosphatase, alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transferase and total bilirubin [TBL]) ≥ 1.5 × upper limit of normal (ULN) on day -1 of period 1.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to first IP administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1 of period 1.
* Subject has any of the following concerns with regard to tuberculosis:

  * History of active tuberculosis
  * Abnormalities detected in a chest X-ray on day -1 of period 1
  * Contact with infectious tuberculous patients
* Subject has any clinically significant abnormality following the physical examination, electrocardiogram (ECG) and protocol-defined clinical laboratory tests at screening or on day -1 of period 1.
* Participant has a mean pulse < 45 bpm, > 99 bpm; mean body temperature < 35.0°C, > 37.5°C; mean systolic blood pressure < 90 mmHg, ≥ 140 mmHg; mean diastolic blood pressure < 40 mmHg, ≥ 90 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes) at screening or on day-1 of period 1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Participant has a mean corrected QT interval using Fridericia's formula (QTcF) of: ≥ 430 msec (for male subjects) ≥ 450 msec (for female subjects) at screening or on day-1 of period 1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Subject has used any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's Wort and traditional Chinese medicine) in the 2 weeks prior to first IP administration, except for occasional use of paracetamol (up to 2 g/day), topical dermatological products, including corticosteroid products, hormonal contraceptives or hormone replacement therapy (HRT).
* Subject has a history of smoking > 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to day -1 of period 1.
* Subject has a history of consuming > 21 units for male subjects or > 14 units for female subjects of alcohol per week within 3 months prior to day -1 of period 1 (note: 1 unit = 10 g pure alcohol, 250 mL of beer [5%], 35 mL of spirits [35%] or 100 mL of wine [12%]) or the subject has a history of alcohol-dependency, drug-dependency, chemical-dependency, or alcohol or drug abuse within 2 years prior to screening or the subject tests positive for alcohol at screening or on day -1 of period 1.
* Subject has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 of period 1 or the subject tests positive for drugs of abuse (amphetamines, benzodiazepines, cannabinoids, cocaine and opiates) at screening or on day -1 of period 1.
* Subject has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1 of period 1.
* Subject has had significant blood loss, donated ≥ 400 mL of whole blood within 90 days, ≥ 200 mL of whole blood within 30 days or donated blood components within 14 days prior to day -1 of period 1 and/or received a transfusion of any blood or blood products within 60 days.
* Subject has a positive serology test for hepatitis A virus antibodies (immunoglobulin M), hepatitis B core antibodies, hepatitis B surface antigen, hepatitis C virus antibodies, human immunodeficiency virus or syphilis at screening.
* Subject is an employee of Astellas, the study-related contract research organizations or the clinical unit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Director, Study Director — Astellas Pharma China, Inc.
Locations (1):
- Site CN86001, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/?pid=178-MA-2294
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14527&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at one site in China.
Pre-assignment Details: Healthy Chinese female and male participants between 18 to 45 years of age, inclusive (at screening), and met all of the inclusion and none of the exclusion criteria were eligible to participate in this study.
Groups:
- Mirabegron 25 mg Fed/Mirabegron 25 mg Fasted: Participants received single dose of 25 milligrams (mg) mirabegron tablet under fed condition orally, on day 1 of period 1 followed by single dose of 25 mg mirabegron tablet under fasted condition orally, on day 1 of period 2. A washout period of 10 days was maintained between the mirabegron administrations in each period.
- Mirabegron 50 mg Fasted/Mirabegron 50 mg Fed: Participants received single dose of 50 mg mirabegron tablet under fasted condition orally, on day 1 of period 1 followed by single dose of 50 mg mirabegron tablet under fed condition orally, on day 1 of period 2. A washout period of 10 days was maintained between the mirabegron administrations in each period.
Period: Period 1 (5 Days)
Arm/Group | Mirabegron 25 mg Fed/Mirabegron 25 mg Fasted | Mirabegron 25 mg Fasted/Mirabegron 25 mg Fed | Mirabegron 50 mg Fed/Mirabegron 50 mg Fasted | Mirabegron 50 mg Fasted/Mirabegron 50 mg Fed
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (10 Days)
Arm/Group | Mirabegron 25 mg Fed/Mirabegron 25 mg Fasted | Mirabegron 25 mg Fasted/Mirabegron 25 mg Fed | Mirabegron 50 mg Fed/Mirabegron 50 mg Fasted | Mirabegron 50 mg Fasted/Mirabegron 50 mg Fed
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 (5 Days)
Arm/Group | Mirabegron 25 mg Fed/Mirabegron 25 mg Fasted | Mirabegron 25 mg Fasted/Mirabegron 25 mg Fed | Mirabegron 50 mg Fed/Mirabegron 50 mg Fasted | Mirabegron 50 mg Fasted/Mirabegron 50 mg Fed
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Mirabegron 25 mg Fed/Mirabegron 25 mg Fasted: Participants received single dose of 25 mg mirabegron tablet under fed condition orally, on day 1 of period 1 followed by single dose of 25 mg mirabegron tablet under fasted condition orally, on day 1 of period 2. A washout period of 10 days was maintained between the mirabegron administrations in each period.
- Total: Total of all reporting groups
Arm/Group | Mirabegron 25 mg Fed/Mirabegron 25 mg Fasted | Mirabegron 25 mg Fasted/Mirabegron 25 mg Fed | Mirabegron 50 mg Fed/Mirabegron 50 mg Fasted | Mirabegron 50 mg Fasted/Mirabegron 50 mg Fed | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.8 (7.8) | 25.0 (4.8) | 26.7 (7.2) | 24.5 (3.7) | 26.0 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4
  Male | 5 | 5 | 5 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 6 | 6 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 6 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under The Concentration-Time Curve (AUC) From The Time of Dosing Extrapolated to Time Infinity (AUCinf) For Mirabegron
Description: AUCinf for mirabegron was reported for the plasma samples collected.
Time Frame: Day 1: predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 72 and 96 hour(s) postdose of each period
Population: The pharmacokinetic analysis set (PKAS) consisted of all participants who received at least 1 dose of investigational product (IP) for which concentration data were available to facilitate derivation of at least 1 primary pharmacokinetic parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter (h*ng/mL)
Groups:
- Mirabegron 25 mg Fed: Participants received single dose of 25 mg mirabegron tablet under fed condition orally, on day 1 of either period 1 or period 2.
- Mirabegron 25 mg Fasted: Participants received single dose of 25 mg mirabegron tablet under fasted condition orally, on day 1 of either period 1 or period 2.
- Mirabegron 50 mg Fed: Participants received single dose of 50 mg mirabegron tablet under fed condition orally, on day 1 of either period 1 or period 2.
- Mirabegron 50 mg Fasted: Participants received single dose of 50 mg mirabegron tablet under fasted condition orally, on day 1 of either period 1 or period 2.
Arm/Group | Mirabegron 25 mg Fed | Mirabegron 25 mg Fasted | Mirabegron 50 mg Fed | Mirabegron 50 mg Fasted
Number analyzed (Participants) | 12 | 12 | 12 | 12
Hour*nanogram per milliliter (h*ng/mL) | 81.8 (37.2) | 143 (39.3) | 263 (26.9) | 429 (36.8)
Statistical Analysis 1: Comparison: Mirabegron 25 mg Fed vs Mirabegron 25 mg Fasted; Assessment based on an analysis of variance (ANOVA) performed on natural log-transformed parameters with food condition and period as a fixed effects and participant as a random effect; Test type: Other; Geomteric Least Squares (LS) Mean Ratio = 57.06, 90% CI 2-sided [46.21 to 70.47] — Ratios and confidence intervals are transformed back to raw scale & values are expressed as percentages
Statistical Analysis 2: Comparison: Mirabegron 50 mg Fed vs Mirabegron 50 mg Fasted; Assessment based on an ANOVA performed on natural log-transformed parameters with food condition and period as a fixed effects and participant as a random effect; Test type: Other; Geometric LSMean Ratio = 61.42, 90% CI 2-sided [52.06 to 72.47] — Ratios and confidence intervals are transformed back to raw scale & values are expressed as percentages

2. Primary Outcome: Area Under The Concentration-Time Curve (AUC) From The Time of Dosing to The Last Measurable Concentration (AUClast) For Mirabegron
Description: AUClast for mirabegron was reported for the plasma samples collected.
Time Frame: Day 1: predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 72 and 96 hour(s) postdose of each period
Population: PKAS Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Mirabegron 25 mg Fed | Mirabegron 25 mg Fasted | Mirabegron 50 mg Fed | Mirabegron 50 mg Fasted
Number analyzed (Participants) | 12 | 12 | 12 | 12
h*ng/mL | 63.3 (36.8) | 119 (40.8) | 218 (25.4) | 369 (39.5)
Statistical Analysis 1: Comparison: Mirabegron 25 mg Fed vs Mirabegron 25 mg Fasted; [analysis description as in outcome 1, analysis 2]; Test type: Other; Geomteric LSMean Ratio = 53.31, 90% CI 2-sided [43.02 to 66.05] — Ratios and confidence intervals are transformed back to raw scale & values are expressed as percentages
Statistical Analysis 2: Comparison: Mirabegron 50 mg Fed vs Mirabegron 50 mg Fasted; [analysis description as in outcome 1, analysis 2]; Test type: Other; Geomteric LSMean Ratio = 59.14, 90% CI 2-sided [49.48 to 70.70] — Ratios and confidence intervals are transformed back to raw scale & values are expressed as percentages

3. Primary Outcome: Maximum Concentration (Cmax) For Mirabegron
Description: Cmax for mirabegron was reported from the plasma samples collected.
Time Frame: Day 1: predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 72 and 96 hour(s) postdose of each period
Population: PKAS Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Mirabegron 25 mg Fed | Mirabegron 25 mg Fasted | Mirabegron 50 mg Fed | Mirabegron 50 mg Fasted
Number analyzed (Participants) | 12 | 12 | 12 | 12
Nanogram per milliliter (ng/mL) | 3.07 (29.9) | 7.88 (82.1) | 15.9 (47.7) | 33.3 (82.7)
Statistical Analysis 1: Comparison: Mirabegron 25 mg Fed vs Mirabegron 25 mg Fasted; [analysis description as in outcome 1, analysis 2]; Test type: Other; Geometric LSMean Ratio = 38.93, 90% CI 2-sided [26.78 to 56.59] — Ratios and confidence intervals are transformed back to raw scale & values are expressed as percentages
Statistical Analysis 2: Comparison: Mirabegron 50 mg Fed vs Mirabegron 50 mg Fasted; [analysis description as in outcome 1, analysis 2]; Test type: Other; Geometric LSMean Ratio = 47.90, 90% CI 2-sided [31.76 to 72.24] — Ratios and confidence intervals are transformed back to raw scale & values are expressed as percentages

4. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a participant administered an study drug, and which does not necessarily have to have a causal relationship with this study drug. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug whether or not considered related to the study drug. An AE is considered "serious" if, in the view of either the investigator or sponsor, the event results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions results in congenital anomaly, or birth defect, requires inpatient hospitalization, other medically important AE. An AE with onset at any time from first dosing until last scheduled procedure was classified as a TEAE.
Time Frame: From date of informed consent signed to end of study (up to 24 days)
Population: The safety analysis set (SAF) consisted of all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Mirabegron 25 mg Fed | Mirabegron 25 mg Fasted | Mirabegron 50 mg Fed | Mirabegron 50 mg Fasted
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  TEAE | 2 | 2 | 2 | 2
  Drug-Related TEAE | 1 | 2 | 2 | 1
  Serious TEAE | 0 | 0 | 0 | 0
  Drug-Related Serious TEAE | 0 | 0 | 0 | 0
  TEAE Leading to Death | 0 | 0 | 0 | 0
  Drug-Related TEAE Leading to Death | 0 | 0 | 0 | 0
  TEAE Leading to Withdrawal of Treatment | 0 | 0 | 0 | 0
  Drug-Related TEAE Leading to Withdrawal of Treatment | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of informed consent signed to end of study (up to 24 days)
Arm/Group | Mirabegron 25 mg Fed | Mirabegron 25 mg Fasted | Mirabegron 50 mg Fed | Mirabegron 50 mg Fasted
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 2/12 | 2/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron 25 mg Fed (N=12) | Mirabegron 25 mg Fasted (N=12) | Mirabegron 50 mg Fed (N=12) | Mirabegron 50 mg Fasted (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT04501640/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT04501640/SAP_001.pdf